CLINICAL TRIAL: NCT04782830
Title: Use of Accelerometer for Quantification of Neurogenic Orthostatic Hypotension Symptoms
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Italo Biaggioni, Professor of Medicine and Pharmacology, Vanderbilt University Medical Center
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: 201219
Record Dates: First submitted 2021-03-01; First posted 2021-03-04 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Orthostatic; Hypotension, Neurogenic; Autonomic Failure; Pure Autonomic Failure; Multiple System Atrophy; Orthostatic; Hypotension, Parkinsonism
Keywords: orthostatic hypotension; autonomic failure; accelerometer; orthostatic symptoms
MeSH Terms: conditions — Hypotension; Pure Autonomic Failure; Multiple System Atrophy; Parkinsonian Disorders; Hypotension, Orthostatic | interventions — Sugars; Midodrine; Atomoxetine Hydrochloride

STUDY DESIGN:
Intervention Model Description: placebo-controlled, double-blind, randomized crossover
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants and outcome assessor will be blinded to the study medications
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- placebo (Experimental): Placebo pill will be taken for 7 days at the same frequency as their regular treatment with either midodrine or atomoxetine.
  Interventions: Device: Accelerometer; Drug: placebo pill
- Standard treatment (Active Comparator): Either midodrine or atomoxetine at their regular dose.
  Interventions: Device: Accelerometer; Drug: Midodrine or atomoxetine pill

INTERVENTIONS:
Device: Accelerometer — A uniaxial accelerometer-based activity monitor (ActivpalTM) will be worn by participants on one of the thighs during the 7 days of the placebo and treatment periods.
  Other Names: ActivpalTM
Drug: placebo pill — Placebo pill will be taken for 7 days at the same frequency as their regular treatment with either midodrine or atomoxetine.
  Other Names: sugar pill
  Arms: placebo
Drug: Midodrine or atomoxetine pill — Either midodrine or atomoxetine at their regular dose.
  Arms: Standard treatment

SUMMARY:
The objective of this study is to find a more objective and accurate way to assess the efficacy of the treatment for neurogenic orthostatic hypotension. For this purpose, the investigators will use an activity monitor to determine the amount of time patients spend in the upright position (standing and walking; upright time) during 1 week of placebo (a pill with no active ingredients) and 1 week of their regular medication for orthostatic hypotension (midodrine or atomoxetine at their usual doses). Total upright time (i.e. tolerance to standing and walking) will be compared between placebo and active treatment to test the hypothesis that it can be used to assess the efficacy of the treatment for orthostatic hypotension and whether this outcome is superior to the assessment of symptoms using validated questionnaires.

DETAILED DESCRIPTION:
Patients with autonomic failure cannot regulate blood pressure properly. Upon standing, their blood pressure drops (i.e. orthostatic hypotension) and may cause symptoms such as lightheadedness, dizziness, changes in vision, weakness, fatigue, trouble concentrating, and shoulder and neck pain. Orthostatic hypotension can be severe and disabling; it can lead to frequent loss of consciousness and falls. These symptoms can make it difficult to perform activities of daily living resulting in significant impairment of the patient's quality of life. Thus, the assessment of orthostatic symptoms using validated questionnaires has been one of the main tools to determine the efficacy of treatment approaches for orthostatic hypotension. However, its usefulness may be limited by several factors including difficulty in the categorization of symptoms and rating of their severity, particularly in patients with some degree of cognitive impairment; the confounding effect of factors not related to orthostatic hypotension on patient's symptoms; difficulty in performing an accurate comparison of the severity of symptoms before and after treatment or between treatments; underestimating symptom burden by not reporting symptoms that are not included in the validated questionnaires or by problems in the patient recall.

The objective of this study is to find a more objective and accurate way to assess the efficacy of the treatment for neurogenic orthostatic hypotension. The main hypothesis is that the quantification of upright time (standing and walking) with an activity monitor would be useful in the assessment of the severity of neurogenic orthostatic hypotension and the efficacy of the treatment for this condition and whether it would be superior to the assessment of symptoms using validated questionnaires.

Patients with autonomic failure and neurogenic orthostatic hypotension on treatment with either midodrine or atomoxetine will be eligible for this study. The study will take place at the participant's home with the assistance of his or her caregiver and frequent oversight from the investigative team. Participants will be studied for two separate weeks, one week with placebo and one week with their regular treatment (midodrine or atomoxetine at their usual doses), with one week in between for washout (the period of using participants' usual medication without any study measurement performed). The order of the study weeks with placebo or regular treatment will be randomized and the study medications will be blinded. On each study week, participants will be asked to wear an activity monitor (Activpal) on one of their thighs to measure the amount of time they spend in the upright posture (walking and standing), number of steps, activity and other characteristics related to the quantity and quality of walking and standing. Participants will be guided to write down the times of their daily activities, such as waking, sleeping, eating, and taking medication. At the end of each study week, the participants will be guided to fill out some questionnaires, and to take blood pressure measurements while lying down, sitting, and standing.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects, age 40-80 years.
* Possible or probable Multiple Systems Atrophy, Pure Autonomic Failure, or Parkinson's disease with neurogenic orthostatic hypotension.
* Neurogenic orthostatic hypotension defined as a ≥ 30 mmHg decrease in systolic blood pressure within 3 minutes of standing associated with impaired autonomic reflexes determined by autonomic testing in the absence of other identifiable causes.
* Patients on treatment for neurogenic orthostatic hypotension with either midodrine or atomoxetine, who have experienced some improvement in their orthostatic symptoms, but still remain symptomatic (Orthostatic hypotension symptom assessment [OHSA] score of 1 to 5 while on medication).
* Patients who are able to stay with their caregiver during study participation.
* Able and willing to provide informed consent.

Exclusion Criteria:

* Bedridden, physically disabled, or unable to walk.
* Patients with Orthostatic hypotension symptom assessment (OHSA) score ≥ 6, or orthostatic systolic blood pressure drop ≥ 30 mmHg on their regular treatment.
* Patients taking more than one medication for the treatment of neurogenic orthostatic hypotension (concomitant use of pyridostigmine or fludrocortisone are accepted).
* Pregnancy
* Systemic illnesses known to produce autonomic neuropathy, including but not limited to diabetes mellitus, amyloidosis, monoclonal gammopathies, and autoimmune neuropathies.
* Clinically unstable coronary artery disease (recurrent angina despite medical therapy), or major cardiovascular or neurological event in the past 6 months (myocardial infarction, stroke).
* Concomitant use of anticoagulants.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Estimated)
Dates: Start 2021-02-05 (Actual); Primary Completion 2027-06-01 (Estimated); Study Completion 2027-10-01 (Estimated)

PRIMARY OUTCOMES:
Total standing time measured by an accelerometer | 7 days of the treatment or placebo period
  The percentage of total standing time during the treatment or placebo period will be measured by an accelerometer (Activpal) placed on one of the patient's thighs. The accelerometer quantifies the length of time spent in the upright and seated or supine positions.
Orthostatic symptoms | 7 days of treatment or placebo period
  Orthostatic symptoms measured by the Orthostatic Hypotension Questionnaire (OHQ). The questionnaire is divided into two parts: Part I, Symptom Assessment (OHSA), consisted of six questions, each rating the intensity of one characteristic symptom of OH: 1) Dizziness, lightheadedness, feeling faint, or feeling like you might blackout; 2) Blurring, seeing spots or tunnel vision; 3) Generalized weakness; 4) Fatigue; 5) Trouble concentrating; 6) Head/neck discomfort; and Part II, Daily Activity Scale (OHDAS), consisted of four questions that assessed the impact of neurogenic OH symptoms on daily activities. The recall period is ''over the past week''. The items are scored on an 11-point scale from 0 to 10, with 0 indicating no symptoms/no interference and 10 indicating the worst possible symptoms/complete interference, and the option of selecting ''cannot be done for other reasons''. The composite OHQ score is calculated by averaging the OHSAS and the OHDAS.

SECONDARY OUTCOMES:
Total number of steps measured by an accelerometer | 7 days of treatment or placebo period
  Number of steps during the treatment or placebo period will be measured by an accelerometer (Activpal) placed on one of the patient's thighs
Total walking time measured by an accelerometer | 7 days of treatment or placebo period
  Total walking time during the treatment or placebo period will be measured by an accelerometer (Activpal) placed on one of the patient's thighs. The accelerometer quantifies the length of time spent walking, standing still, and sitting or lying down.

CONTACTS AND LOCATIONS:
Overall Officials: Italo Biaggioni, MD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Autonomic Dysfunction Center/ Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No